CLINICAL TRIAL: NCT02917499
Title: Efficacy and Safety of TMS and Deep TMS Treatment for Psychiatric and Neurological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sveti Ivan Psychiatric Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMS
Record Dates: First submitted 2016-09-14; First posted 2016-09-28 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Mood Disorders
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- TMS (Experimental): The experimental group will be treated with transcranial magnetic stimulation for 4 weeks.
  Interventions: Device: TMS
- noTMS (No Intervention): The control (no intervention) group will be treated as usual (with pharmacotherapy). These patients will receive TMS treatment after data collection is ended.

INTERVENTIONS:
Device: TMS — Transcranial magnetic stimulation
  Arms: TMS

SUMMARY:
The goal of this study is to examine the efficacy and safety of transcranial magnetic stimulation (TMS) and deep TMS (dTMS) for treatment of different psychiatric and neurological disorders. Subjects will be randomized into two groups: experimental (treated with pharmacotherapy and TMS) and control group (treated only with pharmacotherapy). They and their clinicians will complete a battery of instruments that measure relevant symptoms, global functioning and quality of life. The first measurement will be done after the inclusion and before treatment. The second measurement will be made immediately after the end of treatment (after 4 weeks). The other measurements (follow-up) will be made after 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed psychiatric or neurological disorder, duration of disorder for at least 5 years, inpatients or outpatients treated in Psychiatric hospital Sveti Ivan

Exclusion Criteria:

* suicidality, psychosis, alcohol addiction, unable to complete the questionnaires

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
the proportion of patients who experienced complete remission of the disease | up to six months
  Measurement points: immediately after the end of treatment, and follow-up after 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- PB Sveti Ivan, Zagreb, Croatia

REFERENCES:
- [Derived] Filipcic I, Simunovic Filipcic I, Milovac Z, Sucic S, Gajsak T, Ivezic E, Basic S, Bajic Z, Heilig M. Efficacy of repetitive transcranial magnetic stimulation using a figure-8-coil or an H1-Coil in treatment of major depressive disorder; A randomized clinical trial. J Psychiatr Res. 2019 Jul;114:113-119. doi: 10.1016/j.jpsychires.2019.04.020. Epub 2019 Apr 26. PMID 31059991